CLINICAL TRIAL: NCT06201910
Title: Retrospective Evaluation of Peripartum Blood Loss and Postpartum Anaemia With Respect to Fetal Macrosomia and Gemini
Brief Title: Evaluation of Peripartum Blood Loss and Postpartum Anaemia in Macrosomia & Gemini
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Other Study IDs: 2023-1405
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-03

CONDITIONS: Bloodloss in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Controll: Pregnant women without uterine dilation due to a twin pregnancy or a macrosomic singleton
  Interventions: Other: Observation of Blood loss
- Gemini: Pregnant women with uterine dilation due to a twin pregnancy
  Interventions: Other: Observation of Blood loss
- Makrosome: Pregnant women with uterine dilation due to a macrosomic singleton
  Interventions: Other: Observation of Blood loss

INTERVENTIONS:
Other: Observation of Blood loss — Retrospetive observation of bloodloss and RBC transfusions.

SUMMARY:
Anaemia in pregnant women occurs at a haemoglobin (Hb) concentration <11 g/dL and treatment is essential to prevent increased maternal morbidity, fetal morbidity and mortality. Studies show a distinct risk of haemorrhage in pregnant women due to increased uterine dilatation, due to twins or macrosomic singletons. Currently, prepartum anaemia management, the influence of anaemia and the administration of foreign blood concentrates are insufficiently studied. The investigators intend to conduct a monocentric retrospective analysis of this subcohort.

DETAILED DESCRIPTION:
Patient blood management is essentially based on three pillars, and a meta-analysis has already shown that consistent use can reduce transfusions and mortality. The WHO defines anaemia in pregnant patients as a haemoglobin (Hb) concentration <11 g/dl.

Treatment of iron deficiency anaemia is essential because data show that iron deficiency anaemia is associated with increased maternal morbidity, fetal morbidity and mortality. Studies show a separate risk of bleeding in pregnant women due to increased uterine prolapse, for example in twin pregnancies or macrosomic singletons. At present, the prepartum anaemia management of patients, the influence of anaemia and the administration of foreign blood concentrates are insufficiently studied, which the investigators intend to investigate.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy

Exclusion Criteria:

* pre-existing coagulation disorder

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with or without twin pregnancies or macrosomere singletons
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Bloodloss | Within the first 24 hours after delivery
  Blood loss measured by haemoglobin value

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Goethe University, Frankfurt am Main, Hesse

IPD SHARING:
Plan to Share IPD: No